CLINICAL TRIAL: NCT03597243
Title: Cash Transfer to Adolescent Girls and Young Women to Reduce Sexual Risk Behaviour - an Impact Evaluation
Brief Title: Cash Transfer to Adolescent Girls and Young Women to Reduce Sexual Risk Behavior - an Impact Evaluation
Acronym: CARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Principal Investigator, Mwita Wambura, Principal Research Scientist, National Institute for Medical Research, Tanzania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16.01.CT
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: HIV/AIDS; HSV-2 Infection
Keywords: Cash transfer; HIV; adolescent girls; Tanzania
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Two arms parallel cluster randomized trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): AGYW in the standard Sauti cash transfer (Arm I) will receive unconditional cash transfer (UCT) in the presence of behavioral and biomedical interventions in quarterly installments of 70,000 TSH. The first installment will take place after completion of 10 hours of BCC sessions and the AGYW has registered into CTP.
  Interventions: Other: Cash Transfer
- Control (No Intervention): AGYW in the control group (Arm II) will not receive cash payment but will receive behavioral and biomedical interventions. The behavioral and biomedical interventions are provided by Sauti program to all project beneficiaries.

INTERVENTIONS:
Other: Cash Transfer — Girls enrolled receive a quarterly direct cash transfer of a total of 70,000 Tshs (30 USD) quarterly through mobile phone based cash transfer over a period of two years, for which they will receive mobile phones and SIM cards form the program.
  Arms: Intervention

SUMMARY:
Vulnerability to HIV infection in Adolescent Girls and Young Women (AGYW) is mainly influenced by structural factors which mediate through sexual risk behavior. The Sauti program as implementing partner of the DREAMS initiative will provide unconditional cash transfer on quarterly basis to vulnerable AGYW in selected districts of Tanzania. The CARE study will evaluate the impact of this activity through a cluster randomised controlled trial that involves quantitative and qualitative research techniques. The study will inform policy makers on the impact of Cash transfer programs in AGYW as a tool to reduce vulnerability to HIV infection in Adolescent Girls and Young women.

DETAILED DESCRIPTION:
Vulnerability to HIV infection in Adolescent Girls and Young Women (AGYW) is mainly influenced by structural factors which mediate through sexual risk behaviour. Poverty and few alternative opportunities to generate income make AGYW prone to compensated and often inter-generational and unprotected sex.

The Sauti program as implementing partner of the DREAMS initiative will provide unconditional cash transfer on quarterly basis to vulnerable AGYW in selected districts of Tanzania. The CARE study will evaluate the impact of this activity through a cluster randomised controlled trial that involves quantitative and qualitative research techniques.

Cash transfer interacts with structural factors influencing sexual risk behavior in AGYW, providing alternative source to solve their social and economic needs and hence reducing the pressure to engage in compensated and unprotected sex which further reduces the risk of HSV-2 and HIV acquisition at the population level.

The proposed study (CARE study) is two parallel arms cluster-randomized controlled trial implemented in 3120 adolescent girls and young women (AGYW) aged 15-23 years followed up for 18 months. Participants in randomized clusters will receive a quarterly cash transfer payment through mobile money on their cellular phones in Arm I (Unconditional Cash Transfer) while Arm II will not receive cash transfer payments (Control). The study will be conducted in Kahama Town Council, Ushetu and Msalala District Councils in Shinyanga region in mainland Tanzania.

CARE study will enrol AGYW aged 15-23 years in 3 districts of Tanzania namely Msalala district, Ushetu district and Kahama town council in Shinyanga region. Villages in these areas will be eligible in the trial if they are:

i) Sauti intervention villages receiving cash transfer or control villages ii) with at least 70 AGYW according to the household survey

AGYW found to be HIV and HSV-2 positive at baseline will not be excluded from the study because: 1) excluding them is likely to disclose their HIV or HSV-2 serostatus to the community and therefore expose them to stigma and other social harm; 2) Recruiting them is likely to increase their linkage to care and treatment and also likely to increase ART adherence; 3) They will participate in the interview and information collected will contribute to the study behavioural outcomes (reporting of compensated sex and inter-generational sex)

Up to 3120 participants (1560 participants per arm) will be screened and up to 3060 enrolled. This sample size will achieve 80% power to detect a 35% reduction of HSV-2 incidence between intervention and the control arms and this sample size is also enough to detect a difference in HIV prevalence between the groups of 35% between the intervention and control arms.

Control: No cash transfer.

Intervention: unconditional cash transfer (UCT) in quarterly instalments of 70,000 TSH. The first instalment will take place after completion of 10 hours of BCC sessions and the AGYW has registered into CTP.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent girls and young women aged 15-23 years.
* Graduated from ten hours of Sauti's BCC sessions.
* Resident of the village of recruitment
* Registered into Cash Transfer Program (CTP) (applicable in the CTP areas only).
* Currently out of school (currently not enrolled in primary, secondary or tertiary education. Either they have never been to school or have dropped out of school for at least a month at time of study enrolment) as documented through a previous household survey of the CT Program (Girls roster).
* Willing and able to give voluntary, informed consent/assent to all study procedures including HIV and HSV-2 testing and receive test results.
* (If <18 years) guardian of the minor AGYW is willing to consent for the study procedures except for emancipated minors (i.e. minors who are married, have given birth or demonstrating full independence e.g. living alone or heading the household).

Exclusion Criteria:

* Not willing or able to consent or assent to the study, in case of minor, no consent from guardian. All minors will require guardian consent except for emancipated minors.
* AGYW not willing to test for HIV or HSV-2 or to receive test results.

Ages: 15 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3120 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-07-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
HSV-2 Incidence | 18 months of follow-up
  Proportion of HSV-2 negative girls who are still free of HSV-2 across the two arms

SECONDARY OUTCOMES:
HIV prevalence | 18 months of follow-up
  HIV prevalence will be assessed by comparing the intervention arm against the control
reporting of compensated sex | 18 months of follow-up
  Proportion of girls reporting compensated sex across the two arms
reporting of intergenerational sexual partnerships | 18 months of follow-up
  Proportion of girls reporting intergenerational sexual partnerships across the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Mwita Wambura, PhD, Principal Investigator — NIMR Mwanza
Locations (1):
- Shinyanga region, Kahama, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
As part of the open data policy, all data emanating from this study will be shared with other researchers
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD will shared during study closure
Access Criteria: Will be determined by the funder and sponsor

REFERENCES:
- [Derived] Kuringe E, Christensen A, Materu J, Drake M, Majani E, Casalini C, Mjungu D, Mbita G, Kalage E, Komba A, Nyato D, Nnko S, Shao A, Changalucha J, Wambura M. Effectiveness of Cash Transfer Delivered Along With Combination HIV Prevention Interventions in Reducing the Risky Sexual Behavior of Adolescent Girls and Young Women in Tanzania: Cluster Randomized Controlled Trial. JMIR Public Health Surveill. 2022 Sep 19;8(9):e30372. doi: 10.2196/30372. PMID 36121686
- [Derived] Wambura M, Drake M, Kuringe E, Majani E, Nyato D, Casalini C, Materu J, Mjungu D, Nnko S, Mbita G, Kalage E, Shao A, Changalucha J, Komba A. Cash Transfer to Adolescent Girls and Young Women to Reduce Sexual Risk Behavior (CARE): Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2019 Dec 20;8(12):e14696. doi: 10.2196/14696. PMID 31859686
- [Derived] Nyato D, Materu J, Kuringe E, Zoungrana J, Mjungu D, Lemwayi R, Majani E, Mtenga B, Nnko S, Munisi G, Shao A, Wambura M, Changalucha J, Drake M, Komba A. Prevalence and correlates of partner violence among adolescent girls and young women: Evidence from baseline data of a cluster randomised trial in Tanzania. PLoS One. 2019 Oct 8;14(10):e0222950. doi: 10.1371/journal.pone.0222950. eCollection 2019. PMID 31593577